CLINICAL TRIAL: NCT00541346
Title: Phase III Study of Autism Co-Morbid for Attention Deficit Hyperactivity Disorder
Brief Title: A Pilot Study of Daytrana TM in Children With Autism Co-Morbid for Attention Deficit Hyperactivity Disorder (ADHD) Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Mark L. Wolraich, M.D. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD485-420-Lock
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2013-12

CONDITIONS: Autism; Attention Deficit Hyperactivity Disorder
Keywords: Autism; Autism Spectrum Disorders; ADHD
MeSH Terms: conditions — Autistic Disorder; Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Methylphenidate Transdermal System (Experimental): 10mg for one week, with weekly stepwise increases to 15mg, 20mg, and 30mg for additional 7 weeks, if symptom reports remained elevated. Titration decreased one stepwise dosage
  Interventions: Drug: Methylphenidate Transdermal System

INTERVENTIONS:
Drug: Methylphenidate Transdermal System — 10mg for one week, with weekly stepwise increases to 15mg, 20mg, and 30mg for additional 7 weeks, if symptom reports remained elevated. Titration decreased one stepwise dosage
  Other Names: Daytrana, MethylPatch, MTS

SUMMARY:
This is an open-label study of the efficacy of Daytrana (methylphenidate transdermal system) for the treatment of attention and behavioral symptoms in children with Autism Spectrum Disorders. Twenty patients will be enrolled and treated with 10-30 mg of Daytrana for a total of eight weeks. Changes in core hyperactivity, impulsivity, and inattention symptoms, autism spectrum symptoms and functional outcomes will be assessed. Acceptability of the transdermal route of administration in this population will also be assessed.

The researchers hypothesize that Daytrana is a safe and effective medication for children with Autism Spectrum Disorders who have symptoms of inattention, hyperactivity and impulsivity.

DETAILED DESCRIPTION:
The design will be an open-label trial of eight weeks duration with 20 children with Autism co-morbid for ADHD. The subjects will receive 7 days of 10 mg of Daytrana. The children will be seen weekly for assessment for 4 weeks then every two weeks until the eight week period is complete. After each week of treatment, response will be reassessed and the dose will be increased stepwise to 15 mg, 20 mg, 30 mg unless there are excessive side effects, in which case, the dose will be reduced to the previous dose or the patch wear time may be revised.

ELIGIBILITY:
Inclusion Criteria:

* Between 6 and 11 years
* Autism Spectrum Disorder
* Attention Deficit Hyperactivity Disorder
* Stimulant medication-free at study entry
* No clinically significant abnormalities that preclude safe participation
* Sufficient developmental level (~3 yrs)
* Able to keep appointments
* Able to communicate effectively
* Teacher cooperation

Exclusion Criteria:

* Received an investigational medication in the previous 30 days
* Current medication treatment is effective and well-tolerated
* Medical conditions that affect patient safety
* MAOIs within one month
* Hypertension
* Bipolar disorder or psychosis
* Anticonvulsants
* Psychotropic medication or health food supplement
* Tourette Disorder
* Seizure disorder
* Neurological condition
* Structural heart disease

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2007-09; Primary Completion 2009-05 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Lock, M.D., Principal Investigator — OU Child Study Center; Mark L Wolraich, M.D., Study Director — OU Child Study Center
Locations (1):
- OU Child Study Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Abanilla PK, Hannahs GA, Wechsler R, Silva RR. The use of psychostimulants in pervasive developmental disorders. Psychiatr Q. 2005 Fall;76(3):271-81. doi: 10.1007/s11126-005-2980-7. PMID 16080422

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 enrolled Study Start Date: September, 2007 Study Completion Date:May, 2009 Seen at OU Physician's Child Study Center.
Groups:
- Methylphenidate Transdermal System: 10mg for one week, with weekly stepwise increases to 15mg, 20mg, and 30mg for additional 7 weeks, if symptom reports remained elevated. Titration decreased one stepwise dosage when significant side-effects were present.
Period: Baseline
Arm/Group | Methylphenidate Transdermal System
Started | 16
Completed | 16
Not Completed | 0
Period: Follow-up
Arm/Group | Methylphenidate Transdermal System
Started | 16
Completed | 15
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Methylphenidate Transdermal System
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.83 (1.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Attention Deficit Hyperactivity Disorder Rating Scale - IV (ADHD-RS-IV) Total Score From Baseline to 8-week Follow-up Visit
Description: This instrument is a parent rating scale used to assess the frequency of ADHD symptoms based on DSM-IV criteria. Raw scores range from 0-54. Higher scores indicate a higher frequency of ADHD symptoms. Raw scores were used in the analyses described below.
Time Frame: Baseline, 8 weeks
Population: Intention to Treat (ITT). Bayesian posterior-predictive imputation of the 8th-week follow-up assessment was used to handle missing data for a single drop-out participant who left the study after a 2nd follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate Transdermal System
Number analyzed (Participants) | 16
units on a scale
  Baseline: ADHD-RS-IV Total Score | 39.9 (7.7)
  Follow-Up: ADHD-RS-IV Total Score | 13.8 (9.0)
Statistical Analysis 1: Comparison: Methylphenidate Transdermal System; Random intercept growth curves were fit to all outcome data, including intermediate assessments. A Bayesian posterior-predictive mean change score and its associated 95% credible interval were estimated using the MCMC Gibbs sampler with non-informative priors. Models included linear and quadratic dose effects, effect for compliance, baseline Life Participation Scale (LPS) effect, LPS by compliance interaction, a functional time component, and interaction between LPS and time; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Posterior-Predictive Probability of Mean Change (Pre-Post) Score at or Below Zero; Bayesian random intercept model; Bayesian Mean Change Score = 26.3, 95% CI 2-sided [19.6 to 33.1] — The confidence interval listed is a Bayesian credible interval which represents the probabilistic likelihood that the population mean change falls within these bounds

2. Secondary Outcome: Change in Aberrant Behavior Checklist (ABC) Hyperactivity Scores From Baseline to 8-week Follow-up Visit
Description: The ABC is a behavior rating scale administered by the clinician which is designed to measure behavior changes brought about by drug treatment effects. 16 of these items comprise the hyperactivity, noncompliance factor. Each item is scored on a 3 point scale where 0 indicates the behavior is not a problem and 3 indicates the behavior problem is severe in degree. The minimum score on this factor is 0 (no behavior problems) while the maximum score is 48 ( severe behavior problems).
Time Frame: Baseline, 8 weeks
Population: Intention to Treat (ITT). Bayesian posterior-predictive imputation of the 8th-week assessment was used to handle missing data for a single drop-out participant who left the study after the 2nd follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate Transdermal System
Number analyzed (Participants) | 16
units on a scale
  Baseline: ABC HYPERACTIVITY | 34.1 (8.3)
  Follow-up: ABC HYPERACTIVITY | 11.3 (8.4)
Statistical Analysis 1: Comparison: Methylphenidate Transdermal System; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Posterior-Predictive Probability of Mean Change Score (Pre-Post) at or Below Zero; Bayesian random intercept model; Bayesian Mean Change Score = 23.1, 95% CI 2-sided [16.9 to 29.3] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change in Aberrant Behavior Checklist (ABC) Irritability Scores From Baseline to 8-week Follow-up Visit
Description: The ABC is a behavior rating scale administered by the clinician which is designed to measure behavior changes brought about by drug treatment effects. 15 of these items comprise the irritability/agitation/crying factor. Each item is scored on a 3 point scale where 0 indicates the behavior is not a problem and 3 indicates the behavior problem is severe in degree. The minimum score on this factor is 0 (no behavior problems) while the maximum score is 45 ( severe behavior problems).
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate Transdermal System
Number analyzed (Participants) | 16
units on a scale
  Baseline: ABC Irritability | 19.8 (9.6)
  Follow-up: ABC Irritability | 9.1 (6.5)
Statistical Analysis 1: Comparison: Methylphenidate Transdermal System; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Posterior-Predictive Probability of Mean Change Score (Pre-Post) at or Below Zero; Bayesian random intercept model; Bayesian Mean Change Score = 10.9, 95% CI 2-sided [5.4 to 16.8]

4. Secondary Outcome: Change in Aberrant Behavior Checklist (ABC) Lethargy Scores From Baseline to 8-week Follow-up Visit
Description: The ABC is a behavior rating scale administered by the clinician which is designed to measure behavior changes brought about by drug treatment effects. 16 of these items comprise the lethargy/social withdrawal factor. Each item is scored on a 3 point scale where 0 indicates the behavior is not a problem and 3 indicates the behavior problem is severe in degree. The minimum score on this factor is 0 (no behavior problems) while the maximum score is 48 ( severe behavior problems).
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate Transdermal System
Number analyzed (Participants) | 16
units on a scale
  Baseline: ABC Lethargy | 11.3 (4.9)
  Follow-up: ABC Lethargy | 4.5 (3.6)
Statistical Analysis 1: Comparison: Methylphenidate Transdermal System; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Posterior-Predictive Probability of Mean Change Score (Pre-Post) at or Below Zero; Bayesian random intercept model; Bayesian Mean Change Score = 7.2, 95% CI 2-sided [3.3 to 11.1] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change in Aberrant Behavior Checklist (ABC) Stereotypy Scores From Baseline to 8-week Follow-up Visit
Description: The ABC is a behavior rating scale administered by the clinician which is designed to measure behavior changes brought about by drug treatment effects. 7 of these items comprise the stereotypic behavior factor. Each item is scored on a 3 point scale where 0 indicates the behavior is not a problem and 3 indicates the behavior problem is severe in degree. The minimum score on this factor is 0 (no behavior problems) while the maximum score is 21 ( severe behavior problems).
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate Transdermal System
Number analyzed (Participants) | 16
units on a scale
  Baseline: ABC Stereotypy | 5.6 (5.4)
  Follow-up: ABC Stereotypy | 1.3 (2.3)
Statistical Analysis 1: Comparison: Methylphenidate Transdermal System; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis — Posterior-Predictive Probability of Mean Change Score (Pre-Post) at or Below Zero; Bayesian random intercept model; Bayesian Mean Change Score = 4.1, 95% CI [1.2 to 6.9] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change in Aberrant Behavior Checklist (ABC) Inappropriate Speech Scores From Baseline to 8-week Follow-up Visit
Description: The ABC is a behavior rating scale administered by the clinician which is designed to measure behavior changes brought about by drug treatment effects. 4 of these items comprise the lethargy/social withdrawal factor. Each item is scored on a 3 point scale where 0 indicates the behavior is not a problem and 3 indicates the behavior problem is severe in degree. The minimum score on this factor is 0 (no behavior problems) while the maximum is 12 ( severe behavior problems).
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate Transdermal System
Number analyzed (Participants) | 16
units on a scale
  Baseline: ABC Inappropriate Speech | 5.5 (2.9)
  Follow-up: ABC Inappropriate Speech | 2.1 (2.3)
Statistical Analysis 1: Comparison: Methylphenidate Transdermal System; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Posterior-Predictive Probability of Mean Change Score (Pre-Post) at or Below Zero; Bayesian random intercept model; Bayesian random intercept model. = 3.5, 95% CI 2-sided [1.8 to 5.2] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change in Lifetime Participation Scale (LPS) Total Scores From Baseline to 8-week Follow-up Visit
Description: The LPS was developed to capture treatment-related improvements in adaptive functioning including quality of life, social development, and emotion regulation. There are 24 items scored using a 4-point Likert frequency scale (0=Never or Seldom, 1=Sometimes, 2=Often, 3=Very Often). A summed scale score (possible range of 0 to 72) was used in the analyses described below. Higher scores indicate more adaptive functioning.
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate Transdermal System
Number analyzed (Participants) | 16
units on a scale
  Baseline: LPS Total | 26.6 (9.0)
  Follow-up: LPS Total | 39.9 (12.2)
Statistical Analysis 1: Comparison: Methylphenidate Transdermal System; Random intercept growth curves were fit to all outcome data. A Bayesian posterior-predictive mean change score and its associated 95% credible interval were estimated using the MCMC Gibbs sampler with non-informative priors. Models included linear dose and time effects; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Posterior-Predictive Probability of Mean Change Score (Pre-Post) at or Above Zero; Bayesian random intercept model; Bayesian Mean Change Score = -10.9, 95% CI 2-sided [-16.8 to -5.4] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change in Family III General Scale Summed Score From Baseline to 8-week Follow-up Visit
Description: The Family Assessment measure is a self-report instrument that provides quantitative indices of family strengths and weaknesses. Each items is rated 0 (strongly agree) to 3 (strongly disagree). The General scale produces seven subscales: task accomplishment, role performance, communication, affective expression, involvement, control and values and norms. The minimum score for each subscale is 0 while the maximum score is 15. Higher raw scores indicate a higher number of family problems reported. A total summed score of all scale scores was used in the analyses described below. The possible range of this total score was 0 to 105. Like the subscales, higher values for this total summed score indicate a higher number of family problems reported.
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate Transdermal System
Number analyzed (Participants) | 16
units on a scale
  Baseline: FAM-III Overall | 55.7 (4.1)
  Follow-up: FAM-III Overall | 53.5 (5.2)
Statistical Analysis 1: Comparison: Methylphenidate Transdermal System; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.21, Mixed Models Analysis — Posterior-Predictive Probability of Mean Change Score (Pre-Post) at or Below Zero; Bayesian random intercept model; Bayesian Mean Change Score = 1.94, 95% CI 2-sided [-2.98 to 6.82] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change in Pediatric Evaluation Disability Inventory (PEDI) Caregiver Assistance: Self-Care From Baseline to 8-week Follow-up Visit
Description: The PEDI Caregiver Assistance measures rate the child's function in three domains: Self-care, Mobility, and Social Function. Items are scored 0 (total, where the child is completely dependent on assistance) to 5 (independent, where no assistance is given or required). Scale scores represent summed item scores within each domain. The Self-Care scale score ranges from 0 to 40. A higher score indicates a higher degree of independence in the self-care area.
Time Frame: Baseline, 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate Transdermal System
Number analyzed (Participants) | 16
units on a scale
  Baseline: PEDI Self-Care | 28.8 (7.0)
  Follow-up: PEDI Self-Care | 32.5 (6.5)
Statistical Analysis 1: Comparison: Methylphenidate Transdermal System; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p > 0.06, Mixed Models Analysis — Posterior-Predictive Probability of Mean Change Score (Pre-Post) at or Above Zero; Bayesian random intercept model; Bayesian Mean Change Score = -3.4, 95% CI 2-sided [-7.9 to 0.80] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Change in Pediatric Evaluation Disability Inventory (PEDI) Social Function From Baseline to 8-week Follow-up Visit
Description: The PEDI Caregiver Assistance measures rate the child's function in three domains: Self-care, Mobility, and Social Function. Items are scored 0 (total, where the child is completely dependent on assistance) to 5 (independent, where no assistance is given or required). Scale scores represent summed item scores within each domain. The Social-Function scale score ranges from 0 to 25. A higher score indicates a higher degree of independence in the Social-Function area.
Time Frame: Baseline, 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate Transdermal System
Number analyzed (Participants) | 16
units on a scale
  Baseline: PEDI Social Function | 9.3 (5.0)
  Follow-up: PEDI Social Function | 14.9 (5.8)
Statistical Analysis 1: Comparison: Methylphenidate Transdermal System; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis — Posterior-Predictive Probability of Mean Change Score (Pre-Post) at or Above Zero; Bayesian random intercept model; Bayesian Mean Change Score = -5.26, 95% CI 2-sided [-9.37 to -1.18] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Change in Attention Deficit Hyperactivity Disorder Rating Scale IV: Teacher Assessment Total Scores From Baseline to 8-week Follow-up Visit
Description: This instrument is a teacher rating scale used to assess the frequency of ADHD symptoms based on DSM-IV criteria. Raw scores range from 0-54. Higher scores indicate a higher frequency of ADHD symptoms. Raw scores were used in the analyses described below.
Time Frame: Baseline, 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate Transdermal System
Number analyzed (Participants) | 12
units on a scale
  Baseline: ADHDRS Teacher Total | 32.6 (8.9)
  Follow-up: ADHDRS Teacher Total | 28.0 (14.4)
Statistical Analysis 1: Comparison: Methylphenidate Transdermal System; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.11, Mixed Models Analysis — Posterior-Predictive Probability of Mean Change Score (Pre-Post) at or Below Zero; Bayesian random intercept model; Bayesian Mean Change Score = 7.6, 95% CI 2-sided [-5.6 to 20.7] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Methylphenidate Transdermal System
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methylphenidate Transdermal System (N=16)
tic (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methylphenidate Transdermal System (N=16)
Headache (Nervous system disorders) | 3
fever (Infections and infestations) | 7
irritability (Psychiatric disorders) | 4
appetite, loss of (Metabolism and nutrition disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
nose, inflammation of (General disorders) | 1
sleeping, difficulty (Psychiatric disorders) | 1
vomiting (Gastrointestinal disorders) | 2
diarrhea (Gastrointestinal disorders) | 2
increased salivation (Gastrointestinal disorders) | 1
blood in stool (Gastrointestinal disorders) | 1
constipation (Gastrointestinal disorders) | 1
eyes bloodshot (Eye disorders) | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1
sore throat (Respiratory, thoracic and mediastinal disorders) | 1
congestion (Respiratory, thoracic and mediastinal disorders) | 1
earache (Ear and labyrinth disorders) | 1
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
enuresis (Psychiatric disorders) | 1
skin, dry (Skin and subcutaneous tissue disorders) | 1
sores under nose (Skin and subcutaneous tissue disorders) | 1
irritation 'burning' application site, patch (Skin and subcutaneous tissue disorders) | 1
hives (Skin and subcutaneous tissue disorders) | 1
less social (Psychiatric disorders) | 1
allergies (Immune system disorders) | 1
itchy eyes (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less